CLINICAL TRIAL: NCT06223464
Title: Evaluation of the Relationship Between Adenomyosis and Elastographic Properties of the Cervix
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Dilara SARIKAYA KURT, Specialist Doctor, Ankara Etlik City Hospital
Other Study IDs: AESH-EK1-2023-630
Record Dates: First submitted 2024-01-13; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Adenomyosis
Keywords: adenomyosis; elastography; cervical
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adenomyosis-Case Group: The study will include those diagnosed with adenomyosis who were evaluated by gynecological examination and ultrasonographic imaging after the application to Etlik City Hospital Gynecology and Obstetrics Clinic, aged 18-45 reproductive period, pregnancy status excluded, without cervical infection, pathology and anomaly, without systemic disease findings and diagnoses, without chronic drug use.
- Healthy patients-Control: The study will include those who have been gynecologically examined and evaluated with ultrasonographic imaging after the application to Etlik City Hospital Gynecology and Obstetrics Clinic, aged 18-45 reproductive period, pregnancy status excluded, without cervical infection, pathology and anomaly, without systemic disease findings and diagnoses, without chronic drug use, without adenomyosis diagnosis.

SUMMARY:
This study aims to evaluate the potential of cervical elastography, a non-invasive method, in the accurate diagnosis and clinical course of adenomyosis. Cervical elastography is an imaging method that measures the elasticity properties of cervical tissue using ultrasound technology. This method may be helpful in providing information about the development and clinical course of adenomyosis.

DETAILED DESCRIPTION:
Adenomyosis is the proliferation of endometrial gland and stroma within the myometrium of the uterus. Its prevalence varies between 10% and 40% in epidemiologic data. It often causes painful menstruation, pelvic pain and other gynecologic symptoms. While adenomyosis may be mild in some patients, it may show infiltrative and severe invasion in others. Advanced cases may be resistant to medical treatment and may affect nearby organs, which makes surgical treatment quite complicated. Therefore, early diagnosis of the disease is important for clinical practice. Global enlargement of the uterus, dysmenorrhea (painful menstruation), menorrhagia, abnormal uterine bleeding and pelvic pain are considered typical clinical symptoms of adenomyosis. However, it should be kept in mind that these symptoms coincide with the histologic diagnosis in a very small proportion of cases, 22% to 65%. The diagnosis and treatment of adenomyosis is complex and therefore there is a need to develop better diagnostic tools and treatment strategies for the management of patients. In this context, new imaging modalities such as cervical elastography may be of potential importance.

Our main hypothesis is that cervical elastography values will be significantly higher in patients with adenomyosis compared to patients without adenomyosis. Our secondary hypothesis is that cervical elastography values will be related to the severity and process of adenomyosis and may be an indicator to predict the symptoms and complications of adenomyosis.

The advantages of Cervical Elastography are the following:

It is non-invasive: Cervical Elastography is performed using ultrasound technology and has no known harm. It stands as a potentially safe method compared to existing invasive tests.

Cost-effective and easy to perform: Cervical Elastography is a procedure performed using existing ultrasound equipment at no separate cost. Therefore, it can be easily performed and repeated in clinical settings.

Fast Results: Cervical Elastography provides fast results by acquiring images in real time. This indicates that cervical elastography can be a valuable diagnostic tool in emergency situations or when rapid decision-making is required.

A potential predictive tool: The results of this study may indicate that the value of cervical elastography is a potential tool for predicting adenomyosis. It may be an important step to develop early diagnosis and treatment strategies to improve health in patients with adenomyosis.

The aim of this study was to compare cervical elastography values between groups of patients with and without adenomyosis and to evaluate the potential of cervical elastography values (quantified in kPa) in the diagnosis of adenomyosis.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 18-45 years of age who volunteered and consented to the reproductive period study
* Patients diagnosed with adenomyosis using MUSA criteria

Exclusion Criteria:

* Pregnancy status
* Pelvic/Cervical infection, pathology and anomalies
* History of cervical surgery
* Diagnosis and findings of systemic disease
* Chronic drug use
* Advanced maternal obesity preventing measurement

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will be included in our study as two case groups with and without the diagnosis of adenomyosis, whose age is 18-45 reproductive period, pregnancy status is excluded, without cervical infection, pathology and anomaly, without systemic disease findings and diagnoses, without chronic drug use, whose gynecological examination was performed and evaluated by ultrasonographic imaging after the application to Etlik City Hospital Gynecology and Obstetrics Clinic. MUSA criteria will be used in the diagnosis of adenomyosis and elastography measurements in kPa will be performed similar to the studies in the literature examples section in the file.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-04-18 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Adenomyosis | 2 months
  MUSA Criteria

SECONDARY OUTCOMES:
Diagnosis of Adenomyosis-Cervical Elastography | 4 months
  Cervical Elastography

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patient data is not open to access due to hospital policy. however, the principal investigator can be reached via e-mail if necessary